CLINICAL TRIAL: NCT04770545
Title: A Phase 3, Open-Label, Multicenter, Extension Study to Evaluate the Long-Term Safety and Efficacy of Pegcetacoplan in Subjects With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: An Extension Study to Evaluate the Long-term Safety and Efficacy of Pegcetacoplan (APL-2) in Subjects With Geographic Atrophy Secondary to AMD
Acronym: GALE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL2-GA-305
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-06

CONDITIONS: Geographic Atrophy Secondary to Age-related Macular Degeneration
MeSH Terms: interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegcetacoplan, 15 mg/100 μL, monthly for up to 36 months (Experimental): Participants from Study APL2-103 (NCT03777332) or those who completed the treatment at Month 24 from either Study APL2-303 (Derby, NCT03525613) or Study APL2-304 (Oaks, NCT03525600) and were administered monthly intravitreal (IVT) pegcetacoplan (15 mg/100 μL) or monthly sham will receive IVT pegcetacoplan (15 mg/100 μL) monthly for up to approximately 36 months.
  Interventions: Drug: PEGCETACOPLAN (APL-2)
- Pegcetacoplan, 15 mg/100 μL, every other month (EOM) for up to 36 months (Experimental): Participants from Study APL2-103 (NCT03777332) or those who completed the treatment at Month 24 from either Study APL2-303 (Derby, NCT03525613) or Study APL2-304 (Oaks, NCT03525600) and were administered every other month (EOM) intravitreal (IVT) pegcetacoplan (15 mg/100 μL) or EOM sham will receive IVT pegcetacoplan (15 mg/100 μL) EOM for up to approximately 36 months.
  Interventions: Drug: PEGCETACOPLAN (APL-2)

INTERVENTIONS:
Drug: PEGCETACOPLAN (APL-2) — Complement (C3) Inhibitor

SUMMARY:
This is a phase 3, open-label, multicenter, extension study to evaluate the long-term safety and efficacy of pegcetacoplan (APL-2) in subjects with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) who participated in Study APL2-103 (NCT03777332) or completed the treatment at Month 24 of either Study APL2-303 (Derby, NCT03525613) or Study APL2-304 (Oaks, NCT03525600).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Ocular-specific inclusion criteria apply to the study eye only.

* Subjects must have participated in APL2-103 (NCT03777332) or completed the treatment at Month 24 of either APL2-303 (Derby, NCT03525613) or APL2-304 (Oaks, NCT03525600).
* For subjects who participated in either the 303 or 304 studies, the condition listed below must also be met for participating in this study.

  * Subjects who did not fully stop study drug treatment, but missed the visit at Month 24, can also participate in the study. However, to participate, subjects must be seen within 60 days from the last day of the period allowed for the 24 months visit in the previous study.
* The eyes of subjects must have transparency to permit visualization of parts inside the eye such as the retina and subjects must be able to look steadily at a provided target allowing the doctor to get good quality pictures from the eye.
* Female subjects must be:

  * Women that cannot have children, or
  * Women who can have children must have a negative result of a blood pregnancy test on the first day of the study visit and agree to use ways to avoid pregnancy during the study and 90 days after the last dose of the study medication.
* Males with female partners who can get pregnant must also agree to use ways to avoid pregnancy and agree not to donate sperm while in the study or until 90 days after administering the last dose of the study medication.
* Agree to participate in the study by signing the consent document providing information about the study; and take part in all tests and assessments as required.

Exclusion Criteria:

Subjects cannot take part in the study if the eye that will be treated during the study currently meets any of the following conditions:

* Participants in APL2 303/304 studies who fully stopped study drug treatment before the visit in month 24 but remain in the study to observe the study medication's safety. Those subjects who temporarily paused study drug treatment are still eligible to participate.
* If, according to your doctor you currently have any disease affecting your eyes that could interfere with your vision, including diseases that affect your retina or macula (the center of the back of your eyes). And, if according to your doctor, the disease in your eyes is benign and does not interfere with the study (e.g. diseases that affects the periphery of the retina), you are also eligible to take part in the study.
* If, according to your doctor you currently have any inflammation/infection in or around your eyes that could prohibit you from receiving an injection inside your eyes.
* If, according to your doctor, any current disease that could directly interfere in your participation in the study or that could make it difficult for you to come to the scheduled visits during the next three yearsover the next 36 months.
* If you have known allergies to fluorescein sodium, a solution that is injected into your body for eye testing; or to pegcetacoplan (the study drug) or any inactive substances in pegcetacoplan solution.
* If you currently are pregnant, breastfeed or have a positive pregnancy test.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of ocular and systemic adverse events | Up to 36 Months

SECONDARY OUTCOMES:
Change from baseline in the total area of GA lesion(s) in the study eye (in mm2) | Up to 36 Months
  The total area of GA lesion(s) in the study eye (in mm2) as assessed by FAF at Month 12, Month 24, and Month 36
Change from baseline in NL-BCVA score (study eye) | Up to 36 Months
  NL-BCVA score as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) chart at Month 12, Month 24, and Month 36
Change from baseline in LL-BCVA score (study eye) | Up to 36 Months
  LL-BCVA score as assessed by ETDRS chart at Month 12, Month 24, and Month 36

CONTACTS AND LOCATIONS:
Locations (174):
- United States (98):
  - Retinal Research Institue, LLC, Phoenix, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Atlantis Eyecare, Huntington Beach, California
  - Jacobs Retina Center, UCSD, La Jolla, California
  - Doheny Eye Center UCLA, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Institute of California Medical Group, Palm Desert, California
  - Byers Eye Institute, Stanford University, Palo Alto, California
  - Retina Consultants San Diego, Poway, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Southwest Retina Research Center, LLC, Durango, Colorado
  - Danbury Eye Physicians & Surgeons, PC, Danbury, Connecticut
  - Retina Group of New England - New London, Waterford, Connecticut
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Pinnacle Research Insitute, Fort Lauderdale, Florida
  - Retina Health Center, Fort Myers, Florida
  - National Opthalmic Research Institute, Fort Myers, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Bascom Palmer Eye Institute at Naples, Naples, Florida
  - Palm Beach Gardens, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Retina Associates of Florida, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Georgia Retina, PC, Marietta, Georgia
  - Gailey Eye Clinic Retina Center, Bloomington, Illinois
  - Northwestern Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina and Vitreous Associates of Kentucky, PSC dba Retina Associates of Kentucky, Lexington, Kentucky
  - The Retina Care Center, Baltimore, Maryland
  - Elman Retina Group, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Center, Hagerstown, Maryland
  - Mid Atlantic Retina Specialist, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - New England Retina Consultants, PC, Springfield, Massachusetts
  - Michigan Medicine Kellogg Eye Center, Ann Arbor, Michigan
  - Associated Retinal Consultants, PC, Grand Rapids, Michigan
  - Associated Retinal Consultants, PC, Traverse City, Michigan
  - Vitreoretinal Surgery, Minneapolis, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of NJ, LLC, Bloomfield, New Jersey
  - NJ Retina, Teaneck, New Jersey
  - NJ Retina, Toms River, New Jersey
  - Vision Research Center Eye Associates of NM, Albuquerque, New Mexico
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Vitreous Retina Macula Consultants of New York, New York, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, PS, Charlotte, North Carolina
  - Duke University, Duke Eye Center, Durham, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - Retina Associates of Cleveland, Inc., Cleveland, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Cole Eye Institute, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Retina Associates of Cleveland, Inc., Youngstown, Ohio
  - Retina Vitreous Center, PLLC, Edmond, Oklahoma
  - Oregon Retina LLP, Eugene, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - Eye Health Northwest, Portland, Oregon
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - AIO Visionary Eye Care, West Mifflin, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Center PLLC, Austin, Texas
  - Brown Retina Institute, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Houston Eye Associates, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Associates of South Texas, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Retina Associates of Utah, PC, Murray, Utah
  - University of Utah - John A. Moran Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - The Retina Group of Washington, Fairfax, Virginia
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Vitreoretinal Associates of Washington, Bellevue, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - Retina Health Center, Madison, Wisconsin
  - Retina-Vitreous Associates Medical Group, Madison, Wisconsin
- Argentina (8):
  - Diagnostico Ocular, Buenos Aires
  - Organizacion Medica de Investigacion (OMI), Buenos Aires
  - Fundacion Zambrano, Buenos Aires
  - Centro Oftalmologico Dr. Charles S.A., Buenos Aires
  - Instituto Oftalmologico de Cordoba, Córdoba
  - OFTAR, Mendoza
  - Microcirujia Ocular Rosario, Rosario
  - Oftalmologos Especialistas, Santa Fe
- Australia (8):
  - Marsden Eye Specialist, Parramatta, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Retina, Sydney, New South Wales
  - The Ashley Centre, Westmead, New South Wales
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Retina and Eye Consultantss, Hurstville
  - Lions Eye Institute, Nedlands
  - Save Sight Institute, Westmead
- IPEPO Instituto Da Visao, São Paulo, Brazil
- Canada (3):
  - Ivey Eye Institute, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Retina Centre of Ottawa, Ottawa, Ontario
- Czechia (5):
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba
  - University hospital Kralovske Vinohrady, Prague
  - AXON Clinical, s.r.o., Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Gemini Eye Clinic, Zlín
- France (14):
  - Centre ophtalmologique Saint-Exupery, Saint-Cyr-sur-Loire, Lyon
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - CHU Dijon, Dijon
  - Clinique du Val d'Ouest, Écully
  - Hopital de la Croix-Rousse, Lyon
  - Centre monticelli Paradis, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - Centre Ophtalmol de l Odeon, Paris
  - Hopital Lariboisiere, Paris
  - CHNO des Quinze-Vingts, Paris
  - Centre Ophtalmo. Image/Laser, Paris
  - Maison Rouge Ophthalmologic Center, Strasbourg
  - CHU de Strasbourg Hopital Civil, Strasbourg
- Germany (12):
  - Universitats-Augenklinik Bonn, Bonn
  - Uniklinik Koln, Cologne
  - University Opthalmology Clinic, Freiburg im Breisgau
  - Uni-medizin Gottingen Augenklinik 3.B1.261, Göttingen
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Augenklinik der LMU Munchen, München
  - Klinikum rechts der Isar, München
  - Augenzentrum am St. Franziskus-Hospital, Münster
  - Universitatsklinikum Regensburg, Münster
  - Universitatsklinikum Munster, Münster
  - STZ Eyetrial, Tübingen
- Israel (4):
  - Assaf ha Rofeh MC, Be’er Ya‘aqov
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - IRCCS San Raffaele, Milan
  - ASST Fatebenefratelli-Sacco Ospedale Luigi Sacco, Milan
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Radboud university medical center Oogheelkunde, Nijmegen
- New Zealand (2):
  - Southern Eye Specialists, Christchurch
  - Hamilton Eye Clinic, Hamilton
- Poland (5):
  - Eye Surgery Center Professor Zagorski, Bydgoszcz
  - Oftalmika Eye Hospital, Bydgoszcz
  - Grupo Laser Vision, Rzeszów
  - Oculomedica Eye Centre, Tarnów
  - UNO-MED Centrum Medyne, Tarnów
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Madrid
  - Instituto Oftalmologico Gomez-Ulla, Santiago de Compostela
- United Kingdom (8):
  - Kings College Hospital NHS Trust, London, London
  - Huddersfield Royal Infirmary, Huddersfield, West Yorkshire
  - St James's University Hospital, Leeds, West Yorkshire
  - Bristol Eye Hospital, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - London Vision Clinic, London
  - Oxford Eye Hospital, Oxford
  - Sunderland Eye Infirmary, Sunderland